CLINICAL TRIAL: NCT00882479
Title: Formalizing a Conceptual Framework of Work Domain Knowledge
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Min Zhu, Program Manager-Research, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-SHIS-09-0047
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Knowledge Representation; Knowledge Modeling

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn the daily activities of nutrition management software users through an improved informed consent process and develop a conceptual model to describe these activities. The investigators will gather information from nutrition management software users, and design and test a new prototype of nutrition management software.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be over 21 years old
2. Subjects must be a student or employee in University of Texas
3. Subjects must be able to read and write in English
4. Subjects must be able to give signed informed consent

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inclusion Criteria:
  1. Subjects must be over 21 years old
  2. Subjects must be a student or employee in University of Texas
  3. Subjects must be able to read and write in English
  4. Subjects must be able to give signed informed consent
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhu, MD, MSC, Principal Investigator — UTHSC-Houston
Locations (1):
- Cognitive Informatics Lab, Houston, Texas, United States